CLINICAL TRIAL: NCT00966979
Title: A Prospective, Post-market, Multi-center Study of the Outcomes of the Triathlon® Partial Knee Resurfacing (PKR) Unicondylar Knee System
Brief Title: Triathlon® Partial Knee Replacement (PKR) Outcomes Study
Acronym: PKR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment goals not being met.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 66
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Osteoarthritis, Post-traumatic arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triathlon PKR (Other): All subjects enrolled will receive the Triathlon PKR device.
  Interventions: Device: Triathlon PKR

INTERVENTIONS:
Device: Triathlon PKR — Triathlon PKR is a unicondylar knee resurfacing system designed to replace a single osteoarthritic compartment of a patient's natural knee.

SUMMARY:
The purpose of this study is to compare the 10-year Knee Society Score (KSS) functional results of the Triathlon PKR Unicondylar Knee to the 10-year Knee Society Score (KSS) functional results of the Triathlon Cruciate Retaining (CR) Total Knee.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or non-pregnant female 21-75 years of age at the time of enrollment.
* The subject requires a primary cemented unicompartmental knee replacement.
* The subject has a diagnosis of osteoarthritis (OA) or posttraumatic arthritis (TA).
* The subject has clinically intact cruciate and collateral ligaments and no ligamentous instability is present.
* The subject has less than 10 degrees of flexion contracture and greater than 90 degrees of flexion.
* The subject's preoperative mechanical alignment is less than 15 degrees of varus and 15 degrees of valgus.
* The subject has signed the Institutional Review Board (IRB) approved study specific Informed Patient Consent Form.
* The subject is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* The subject has inflammatory arthritis or avascular necrosis(AVN).
* The subject is obese, BMI > 35.
* The subject has a history of total or unicompartmental (contralateral compartment and/or patellofemoral joint) reconstruction of the affected joint.
* The subject has a history of anterior cruciate ligament (ACL) reconstruction.
* The subject has had a high distal femoral, or proximal tibial osteotomy.
* The subject has a mental, neuromuscular or neurosensory disorder, which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in post-operative care and/or limit the ability to assess the performance of the device.
* The subject has a systemic or metabolic disorder leading to progressive bone deterioration that the surgeon feels would affect the overall outcome of the study.
* The subject is immunologically suppressed, or is receiving chronic steroids (>30 days duration).
* The subject has a known sensitivity to device materials.
* The subject's bone stock is compromised by disease and/or infection which cannot provide adequate support and/or fixation to the prosthesis.
* The subject's bone stock is compromised by a prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* The subject has an active or suspected latent infection in or about the knee joint.
* The subject is a prisoner.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2023-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. David Heekin, M.D., Principal Investigator — St. Vincent's Medical Center; Marco Tinius, MD, Principal Investigator — Praxisklinik Stollberg; Marco Schiraldi, MD, Principal Investigator — Presidlo Ospedaliero Civile Santi Antonio e Biagio; Brian Aros, MD, Principal Investigator — Mansfield Orthopaedics; Fabio Orozco, MD, Principal Investigator — Rothman Institute; Matthew Phillips, MD, Principal Investigator — Department of Orthopaedic Surgery, Kaleida Health, Buffalo General Hospital; Peter Bonutti, MD, Principal Investigator — Bonutti Clinic; Soren Toksvig-Larsen, MD, Principal Investigator — Hassleholm Sygehus Ortopaedkirurgisk afd.; Brett Greenky, MD, Principal Investigator — Syracuse Orthopedic Specialists; Paul Jacob, MD, Principal Investigator — Oklahoma Sports Science and Orthopaedics
Locations (9):
- United States (6):
  - Heekin Orthopaedic Institute for Research, Inc., Jacksonville, Florida
  - Rothman Institute, Egg Harbor, New Jersey
  - Department of Orthopaedic Surgery, Kaleida Health, Buffalo General Hospital, Buffalo, New York
  - Syracuse Orthopedic Specialists, Syracuse, New York
  - Rothman Institute, Media, Pennsylvania
  - Mansfield Orthopaedics, Morrisville, Vermont
- Praxisklinik Stollberg und Arthro. Zentrum GmbH, Stollberg, Germany
- Presidlo Ospedaliero Civile Santi Antonio e Biagio, Alessandria, Italy
- Hassleholm Sygehus Ortopaedkirurgisk afd. Esplanadgatan, Hässleholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 112 knees in 111 patients that were enrolled in the study (one bilateral case).
Pre-assignment Details: Of the 111 participants enrolled, there were 23 cases that were censored due to not having the study device, surgery canceled or an inclusion exclusion violation. Therefore, 89 knees in 88 participants are followed who did receive the study device and met protocol criteria. Those applicable data are reflected in this record.
Units Other Than Participants: Knees
Groups:
- Triathlon PKR Unicompartmental Knee: All subjects enrolled will receive the Triathlon PKR device.
  Triathlon PKR: Triathlon PKR is a unicondylar knee resurfacing system designed to replace a single osteoarthritic compartment of a patient's natural knee for a primary replacement indication.
Period: Overall Study
Arm/Group | Triathlon PKR Unicompartmental Knee
Started | 111; 112 Knees
Completed | 13; 13 Knees
Not Completed | 98; 99 Knees
Not completed — Death | 1
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 14
Not completed — Adverse Event | 5
Not completed — Sponsor terminated early | 49
Not completed — Censored because surgery not done | 2
Not completed — Censored because study device was not implanted | 14
Not completed — Censored because of Inclusion/exclusion violation | 7

BASELINE CHARACTERISTICS:
Arm/Group | Triathlon PKR
Number analyzed (Participants) | 88
Age, Continuous [Mean (Full Range); unit: years] | 61.83 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 86
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigation of Clinical Performance and Patient Outcome With the Functional Knee Society Score (KSS).
Description: The Knee Society Score (KSS) consists of two distinct sub-scores: one for pain, range of motion, joint stability and alignment (Pain/Motion KSS) and one for distance walked, stair climbing and walking aids (Functional KSS).
  This outcome measure was only for the KSS Function Score at 10-years. The KSS Function score subscale is 0-100, with 100 representing a better outcome. Although the specific scores are not distinguished as "excellent", "good", "fair", or "poor", a higher value represents a better outcome.
Time Frame: 10 years
Population: Due to early study termination the primary outcome was only reached for a minimal number of participants (12) reaching 10 years. These only included prospective cases. No retrospective cases reached the 10-year time interval.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Triathlon PKR Unicompartmental Knee
Number analyzed (Participants) | 12
Number analyzed (Knees) | 12
units on a scale | 98.33 (5.77)

2. Secondary Outcome: 10-years Kaplan Meier Survival Analysis
Description: For the purpose of this study the Kaplan-Meier survival curves are a statistical method to estimate the survival function from lifetime data of a knee replacement after treatment. Survivorship is defined as a percentage of knees free of any component revision for any reason.
Time Frame: 10-years
Population: This primary outcome measure at 10 years is a statistical estimation based on 80 prospective knees as per the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of knees
Units Other Than Participants: Knees
Arm/Group | Triathlon PKR Unicompartmental Knee
Number analyzed (Participants) | 80
Number analyzed (Knees) | 80
percentage of knees | 91.35 [80.12 to 96.37]

ADVERSE EVENTS:
Time Frame: This study required that all operative site adverse events, regardless of seriousness, and serious systemic events, be reported from enrollment to the 10-year postoperative time interval.
Description: The date of occurrence, date diagnosed, type of complication/adverse event and treatment were collected.
Groups:
- Operative Adverse Events: Operative site adverse events are reported by knee because in the case of bilateral participants (this is when one participant has both knees enrolled in the study), an event can occur in one knee, both knees or the same knee at different times and are counted separately for this reason.
- Non-Operative Adverse Events: Non-operative site adverse events are reported by participant.
Arm/Group | Operative Adverse Events | Non-Operative Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/89 | 1/88
Serious Adverse Events (participants affected / at risk) | 11/89 | 20/88
Other Adverse Events (participants affected / at risk) | 26/89 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=89) | Non-Operative Adverse Events (N=88)
Non-operative (Cardiac disorders) | 0/0 (0) | 6 (6)
Non-operative (Gastrointestinal disorders) | 0/0 (0) | 3 (3)
Non-operative (General disorders) | 0/0 (0) | 2 (2)
Operative site (Injury, poisoning and procedural complications) | 1 (1) | 0/0 (0)
Operative site (Musculoskeletal and connective tissue disorders) | 10 (10) | 0/0 (0)
Non-operative (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 4 (4)
Non-operative site (Psychiatric disorders) | 0/0 (0) | 1 (1)
Non-operative (Renal and urinary disorders) | 0/0 (0) | 2 (2)
Non-operative (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
Non-operative (Vascular disorders) | 0/0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative Adverse Events (N=89) | Non-Operative Adverse Events (N=88)
Operative (Musculoskeletal and connective tissue disorders) | 26 (26) | 0 (0)

LIMITATIONS AND CAVEATS:
After 13-years the enrollment goal was not met. This led to a protocol amendment to include retrospective cases. These cases were combined with the initial prospective cases and followed prospectively for the planned observation time. This study does not compare prospective to retrospective cases. The retrospectively enrolled cases were followed prospectively and there were no retrospective cases that reached the 10-year time point, only 12 prospective cases had 10-year data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between Principal Investigators and the Sponsor (or its agents) that requires Investigators to allow Sponsor at least 60 days to review material intended for publications to ensure that confidential information is not disclosed and that the data is accurately represented. The investigators can submit publication proposals prior to the study completion date for Sponsor consideration and for up to 7 years after study completion.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT00966979/Prot_SAP_ICF_000.pdf